CLINICAL TRIAL: NCT01534533
Title: The Effects of Lutein Supplementation on Subclinical Atherosclerosis
Brief Title: Effects of Lutein Supplementation on Subclinical Atherosclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaoming Lin, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NNSFC-30972472; XLin (Registry Identifier: XLin)
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-06

CONDITIONS: Carotid Atherosclerosis; Carotid Intimal Medial Thickness 1
Keywords: early atherosclerosis; serum lutein; serum lycopene; intima-media thickness; arterial stiffness; combined effect
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Intimal Medial Thickness 1; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): early atherosclerosis cases, received starch in hard shell gelatine capsules, once a day
  Interventions: Dietary Supplement: Placebo
- Lutein group (Experimental): early atherosclerosis cases, received 20mg lutein, once a day
  Interventions: Dietary Supplement: Lutein group
- Combination group (Experimental): early atherosclerosis cases, received 20mg lutein plus 20mg lycopene, once a day
  Interventions: Dietary Supplement: Combination group
- Normal lutein control group (Experimental): 20mg lutein for subjects free from atherosclerosis, once a day
  Interventions: Dietary Supplement: Normal lutein control group

INTERVENTIONS:
Dietary Supplement: Placebo — one gelatine capsule containing starch per day, for 12 months
  Arms: Placebo
Dietary Supplement: Lutein group — one gelatine capsule containing 20mg lutein per day, for 12 months
  Arms: Lutein group
Dietary Supplement: Combination group — one gelatine capsule containing 20mg lutein and 20 mg lycopene per day, for 12 months
  Arms: Combination group
Dietary Supplement: Normal lutein control group — subjects without early atherosclerosis, treated with one gelatine capsule containing 20mg lutein per day, for 12 months
  Arms: Normal lutein control group

SUMMARY:
This study is to investigate the possible positive effects of lutein and lycopene supplementation on early atherosclerosis in Beijing.

DETAILED DESCRIPTION:
Atherosclerosis is the primary cause of cardiovascular and cerebrovascular diseases, both of which are the top two causes of death in industrialized countries including China. Lutein was found to be protective against atherosclerosis in some case control studies. However, the intervention on atherosclerosis have not been reported. In the present study, 192 subjects were randomly assigned to four groups treated with different amounts of lutein. The investigators observe the changes of serum lutein concentration by hyper-pressure liquid chromatography (HPLC), and compare the differences of common carotid IMT and arterial stiffness by carotid ultrasonography before and after the intervention. Serum biochemistry indexes including cholesterol (CHO), triglyceride (TG), high density lipoprotein-cholesterol (HDL-C), low density lipoprotein-cholesterol (LDL-C) and glucose (Glu) were measured at 0, 7 and 12 months of treatment by auto-analyzer.

ELIGIBILITY:
Inclusion Criteria:

* early atherosclerosis;
* aged 45 to 68 years;
* Han nationality

Exclusion Criteria:

* history of myocardial infarction,
* stroke,
* revascularization,
* coronary by-pass operation,
* local carotid IMT > 1300μm or supplemental vitamin and/or mineral use for ≥ 4 week before the start of the study

Ages: 45 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Lin, M.M., Principal Investigator — Peking University
Locations (1):
- Haidian District, Beijing, China

REFERENCES:
- [Background] Zou Z, Xu X, Huang Y, Xiao X, Ma L, Sun T, Dong P, Wang X, Lin X. High serum level of lutein may be protective against early atherosclerosis: the Beijing atherosclerosis study. Atherosclerosis. 2011 Dec;219(2):789-93. doi: 10.1016/j.atherosclerosis.2011.08.006. Epub 2011 Aug 10. PMID 21872250

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: starch in hard shell gelatine capsules
- Lutein Group: 20mg lutein per day
- Lutein and Lycopene Group: lutein plus lycopene group
- Normal Lutein Group: subjects without early atherosclerosis
Period: Overall Study
Arm/Group | Placebo | Lutein Group | Lutein and Lycopene Group | Normal Lutein Group
Started | 48 | 48 | 48 | 48
Completed | 40 | 45 | 40 | 44
Not Completed | 8 | 3 | 8 | 4
Not completed — Lost to Follow-up | 3 | 0 | 4 | 3
Not completed — Withdrawal by Subject | 5 | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lutein Group | Lutein and Lycopene Group | Normal Lutein Group | Total
Number analyzed (Participants) | 48 | 48 | 48 | 48 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 44 | 46 | 179
  >=65 years | 3 | 4 | 4 | 2 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 57.4 (5.0) | 57.4 (4.4) | 57.3 (4.9) | 53.8 (5.8) | 56.5 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 28 | 26 | 32 | 116
  Male | 18 | 20 | 22 | 16 | 76
Region of Enrollment [Number; unit: participants]
  China | 48 | 48 | 48 | 48 | 192

OUTCOME MEASURES:

1. Primary Outcome: Table 1 Study Specific Characteristic Part One
Description: The percentage of female, race, hypertenion history, diabetes history, and hyperlipemia history was calculated.
Time Frame: at baseline
Population: We conducted a per protocol analysis of all the subjects who completed the study.
Measure: Number; unit: Percentage of Participants
Groups:
- Placebo (P Group): starch in hard shell gelatine capsules
- Lutein Group (L Group): early atherosclerosis case received 20mg lutein
- Lutein and Lycopene Group (LL Group): received 20mg lutein and 20mg lycopene
- Normal Lutein Control Group (NL Group): subjects free from atherosclerosis received 20mg lutein
Arm/Group | Placebo (P Group) | Lutein Group (L Group) | Lutein and Lycopene Group (LL Group) | Normal Lutein Control Group (NL Group)
Number analyzed (Participants) | 40 | 45 | 40 | 44
Percentage of Participants
  Female | 69.8 | 59.8 | 59.1 | 72.7
  Race (Han people) | 100 | 100 | 100 | 100
  Hypertension history | 63.4 | 57.4 | 56.8 | 20.9
  Diabetes history | 12.2 | 14.9 | 13.6 | 25.6
  Hyperlipemia history | 73.2 | 72.3 | 75.0 | 65.1
Statistical Analysis 1: Comparison: Placebo (P Group) vs Lutein Group (L Group) vs Lutein and Lycopene Group (LL Group); The null hypothesis was "no group difference"; Test type: Superiority or Other; p > 0.05, Chi-squared — The a priori threshold for statistical significance was 0.05 (two sides)

2. Primary Outcome: Table 1 Study Specific Characteristic of Age
Description: the mean and standard deviation of age was calculated in four groups
Time Frame: at baseline
Population: We conducted a per protocol analysis of all the subjects who completed the study.
Measure: Mean (Standard Deviation); unit: years
Groups:
- Combination Group (LL Group): received 20mg lutein and 20mg lycopene
Arm/Group | Placebo (P Group) | Lutein Group (L Group) | Combination Group (LL Group) | Normal Lutein Control Group (NL Group)
Number analyzed (Participants) | 40 | 45 | 40 | 44
years | 57.4 (5.0) | 57.4 (4.4) | 57.3 (4.9) | 53.8 (5.8)
Statistical Analysis 1: Comparison: Placebo (P Group) vs Lutein Group (L Group) vs Combination Group (LL Group); The null hypothesis was "no group difference"; Test type: Superiority or Other; p = 0.992, ANOVA — The a priori threshold for statistical significance was 0.05 (two sides)

3. Primary Outcome: Table 1 Study Specific Characteristic of Body Mass Index (BMI)
Description: the mean and standard deviation of BMI in four groups was calculated
Time Frame: at baseline
Population: We conducted a per protocol analysis of all the subjects who completed the study.
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Placebo (P Group) | Lutein Group (L Group) | Combination Group (LL Group) | Normal Lutein Control Group (NL Group)
Number analyzed (Participants) | 40 | 45 | 40 | 44
Kg/m^2 | 25.3 (2.6) | 25.4 (3.2) | 24.8 (3.2) | 24.1 (2.7)
Statistical Analysis 1: Comparison: Placebo (P Group) vs Lutein Group (L Group) vs Combination Group (LL Group); The null hypothesis was "no group difference"; Test type: Superiority or Other; p = 0.672, ANOVA — The a priori threshold for statistical significance was 0.05 (two sides)

4. Primary Outcome: Table 1 Study Specific Characteristic of Blood Pressure (BP)
Description: systolic BP and diastolic BP in four groups was measure twice between 15minutes
Time Frame: at baseline
Population: We conducted a per protocol analysis of all the subjects who completed the study.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo (P Group) | Lutein Group (L Group) | Lutein and Lycopene Group (LL Group) | Normal Lutein Control Group (NL Group)
Number analyzed (Participants) | 43 | 47 | 44 | 44
mm Hg
  Systolic BP | 129.7 (14.3) | 125.5 (16.4) | 126.0 (15.5) | 117.7 (11.9)
  Diastolic BP | 82.6 (10.6) | 80.5 (9.6) | 80.5 (9.6) | 77.2 (8.1)
Statistical Analysis 1: Comparison: Placebo (P Group) vs Lutein Group (L Group) vs Lutein and Lycopene Group (LL Group); The null hypothesis was "no group difference"; Test type: Superiority or Other; p = 0.402, ANOVA — The a priori threshold for statistical significance was 0.05 (two sides)

5. Primary Outcome: Table 1 Study Specific Characteristic of Serum Carotenoids
Description: serum major carotenoids, including lutein, zeaxanthin, beta-carotene, and lycopene concentration were measured by hyper-pressure liquid chromatography (HPLC)
Time Frame: at baseline
Population: We conducted a per protocol analysis of all the subjects who completed the study.
Measure: Mean (Standard Deviation); unit: μg/ml
Groups:
- Combination Group (LL Group): early atherosclerosis cases received 20mg lutein and 20mg lycopene
Arm/Group | Placebo (P Group) | Lutein Group (L Group) | Combination Group (LL Group) | Normal Lutein Control Group (NL Group)
Number analyzed (Participants) | 40 | 45 | 40 | 44
μg/ml
  Lutein | 0.17 (0.07) | 0.19 (0.14) | 0.20 (0.11) | 0.18 (0.11)
  Zeaxanthin | 0.034 (0.022) | 0.034 (0.018) | 0.035 (0.022) | 0.030 (0.022)
  beta-carotene | 0.087 (0.026) | 0.069 (0.026) | 0.071 (0.031) | 0.058 (0.005)
  Lycopene | 0.106 (0.037) | 0.092 (0.043) | 0.104 (0.074) | 0.098 (0.038)
Statistical Analysis 1: Comparison: Placebo (P Group) vs Lutein Group (L Group) vs Combination Group (LL Group); The null hypothesis was "no group difference"; Test type: Superiority or Other; p = 0.636, ANOVA — The a priori threshold for statistical significance was 0.05 (two sides)

6. Secondary Outcome: Changes of Right Common Carotid Arterial Stiffness Parameter β(R-β) at Baseline and After 12 Months
Description: Arterial stiffness was measured by using a high-resolution B-mode carotid ultrasound with echo-tracking system (Aloka prosound α-10, Aloka Co. Ltd., Tokyo, Japan).
Time Frame: at baseline and after 12 months
Reporting Status: Not Posted, anticipated posting 3333-12

7. Secondary Outcome: Dietary Intake of Energy During the Study Periods
Description: Dietary intake was assessed at baseline and after 12months by using 3 consecutive 24-hour recalls.
Time Frame: at baseline and 12 months
Reporting Status: Not Posted, anticipated posting 3333-12

8. Secondary Outcome: Dietary Intake of Vitamin C,Vitamin E, Lutein Plus Zeaxanthin and Lycopene During the Study Periods
Description: Dietary intake of Vitamin C,Vitamin E, Lutein plus zeaxanthin and Lycopene was assessed at baseline and after 12months by using 3 consecutive 24-hour recalls.
Time Frame: at baseline and 12 months
Reporting Status: Not Posted, anticipated posting 3333-12

ADVERSE EVENTS:
Time Frame: adverse event data were collected in 12months
Arm/Group | Placebo | Lutein Group | Combination Group | Normal Lutein Control Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/45 | 0/40 | 0/44
Other Adverse Events (participants affected / at risk) | 0/40 | 0/45 | 0/40 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes